CLINICAL TRIAL: NCT00761397
Title: Adherence to Swallowing Exercises in Head and Neck Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2008-0360
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Head and Neck Cancer
Keywords: Oropharyngeal cancer; Dysphagic; Swallowing exercises; Swallowing rehabilitative regimens; PREPARE; Patients' Radiation Expectations; Prevention, Adherence, Rehabilitative Exercises
MeSH Terms: conditions — Head and Neck Neoplasms; Oropharyngeal Neoplasms | interventions — Interviews as Topic; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Program Group
  Interventions: Behavioral: Interview; Behavioral: Phone Call; Other: Questionnaire
- Usual Care Group
  Interventions: Other: Brochure; Other: Questionnaire

INTERVENTIONS:
Behavioral: Interview — 15-30 Minute Weekly meeting w/Staff to discuss swallowing exercises
  Groups: Study Program Group
Behavioral: Phone Call — Phone call follow ups for 4 weeks after last radiation treatment
  Groups: Study Program Group
Other: Brochure — Detailed brochure explaining the purpose of the swallowing exercises and a description of how to perform the exercises
  Groups: Usual Care Group
Other: Questionnaire — Day 1 of study, 10 weeks after starting study, & 12 months after starting study

SUMMARY:
The goal of this research study is to help patients complete the swallowing and dental care exercises they are supposed to perform during radiation treatment.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be taught ways to cope with the side effects of radiation as a way to help you do your swallowing exercises during radiation treatment. To find out if the swallowing exercises are being performed, researchers will compare 2 groups of participants.

Study Groups:

You will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups, the Study Program Group or the Usual Care Group. You will have an equal chance of being in either group.

As a part of standard of care, a speech pathologist will teach you how to perform swallowing exercises.

If you are assigned to the Study Program Group, you will complete the following:

* You will meet 1 time a week with study staff during radiation treatment either by phone or in person. These meetings will last between 15 to 30 minutes. During the meetings, you will be asked how many swallowing exercises you have completed during the last week and about any problems you may have had completing the exercises.
* You will receive phone calls for 4 weeks after the last radiation treatment. These phone calls will also last between 15 and 30 minutes. The study staff will ask questions about if you have been doing your exercises and discuss tips to help you continue to do them.
* You will receive a weekly newsletter that has information about ways to cope with any problems you may experience when completing the swallowing exercises.

If you are assigned to the Usual Care Group, you will complete the following:

* The study staff will follow up with you before and during your radiation treatments to make sure that you are scheduled with and have attended your speech pathology appointments. At these appointments, you will be taught how to do the swallowing exercises and given information to help you complete the exercises.
* You will receive a detailed brochure explaining the purpose of the swallowing exercises and a description of how to perform the exercises.
* You will be asked if you would like to participate in another study protocol.

Questionnaires:

Participants in both groups will fill out a questionnaire asking questions about whether or not you have been completing the swallowing and dental exercises and how you have been coping with stress. The questionnaire will also collect information about the disease and demographic information such as age, gender, race, education level, and marital status. This questionnaire will take about 30 minutes to complete each time. You will complete this questionnaire on Day 1, and again 6 weeks, 6 months, 1 year, and 2 years after completing radiation treatment. The second and third questionnaires will be mailed to you along with a stamped envelope for you to return the questionnaires.

Interview:

You will be interviewed. The interview will ask questions about your successful strategies for coping with radiation side effects.

If you disclose through your assessments or discussion that you are having suicidal thoughts or could benefit from antidepressant medication, you may be referred for a consultation with Dr. Alan Valentine, an M. D. Anderson psychiatrist participating in this research study. Study staff will also let your treating doctor and/or regular doctor know about the referral for consultation.

Newsletter:

You will allow the research staff to record any successful strategies for coping with radiation side effects in a written newsletter that will be given to future participants.

Length of Study:

You will remain on study for up to 2 years.

This is an investigational study.

Up to 350 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women are eligible if they a) are predispositioned to receive radiation treatment for oropharyngeal, laryngeal, hypopharyngeal, nasopharyngeal, or an unknown primary cancer with cervical metastases,
2. are stage II-IVB for oropharyngeal and laryngeal
3. are stage I-IVB for hypopharyngeal and nasopharyngeal
4. at least 18 years of age,
5. speak English,
6. are oriented to time, person, and place,
7. and have a Zubrod performance status of 0 to 2.

Exclusion Criteria:

1. have other cancer diagnoses, except non-melanoma skin cancer,
2. had treatment for previous H & N cancer or radiation to the head and neck, or
3. history of previous head and neck surgery (excluding biopsy, tonsillectomy, tracheotomy or selective neck dissection),
4. history of current oropharyngeal dysphagia unrelated to cancer diagnosis (e.g. dysphagia due to underlying neurogenic disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with head and neck cancer who previously had radiation treatment
Sampling Method: Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2008-08-29 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Categorized Adherence Score (e.g., not adherence at all, somewhat adherent, and adherent to all exercises) | Day 1, 10 Weeks, and at 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Eileen H. Shinn, PHD, MS, BA, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org